CLINICAL TRIAL: NCT03055260
Title: Effect of Low Intensity Blood Flow Restriction Training on Lower Extremity Strength and Hypertrophy
Brief Title: Low Intensity Blood Flow Restriction Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Fairview Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1612M02121
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Muscle Mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blood flow restriction cuff (Experimental): This group will receive an active cuff that partially restricts blood flow to the experimental limb.
  Interventions: Device: Blood flow restriction cuff
- Blood Flow restriction Cuff-Placebo (Placebo Comparator): This group will wear a placebo cuff, of which will not restrict blood flow at all.
  Interventions: Device: Blood Flow restriction Cuff-Placebo

INTERVENTIONS:
Device: Blood flow restriction cuff — The intervention is the wearing of a cuff-like band around the affected limb, of which partially restricts blood flow to the limb.
  Arms: Blood flow restriction cuff
Device: Blood Flow restriction Cuff-Placebo — The intervention is the wearing of a cuff-like band around the affected limb, of which partially restricts blood flow to the limb.
  Arms: Blood Flow restriction Cuff-Placebo

SUMMARY:
The particpant will complete baseline testing by measuring subjects' quadriceps muscle thickness (cm) via ultrasound technology, as well as have them complete a one repetition maximum (1RM) test on the leg press machine and an isometric knee extension using a dynamometer - strength measures will be calculated for both right and left legs. After baseline testing, subjects will complete 6 weeks of the testing protocol that will consist of leg press exercises at 30% of their 1RM. Subjects will be randomized to either wear a cuff that partially restricts blood flow to the limb (Study Group), or to wear a cuff that does not restrict blood flow (Control Group). Exercises will be completed 2x/week and will take approximately 10 total minutes (5 for warm up, 5 for testing protocol) per session. After 6 weeks, muscle thickness, leg press 1RM, and quadriceps extension strength will be re-tested and compared to the initial measurements.

DETAILED DESCRIPTION:
Session 1 - baseline testing

* 5-minute warm-up; 1RM calculation for both right and left legs using a supine leg press machine; isometric quadriceps strength measurement using a dynamometer; muscle thickness measurements of both right and left quadriceps muscle using ultrasound technology.
* After day 1 testing; randomly allocate subjects to either control group or experimental group

Sessions 2-13 - 6 weeks of exercise protocol, 2x/per week

Both the experimental and control groups will complete the same protocol for the entirety of the study:

* 5- minute warm up
* Using a single-leg press exercise machine: Subjects complete the testing protocol with either partial blood flow restriction (cuff inflated to 100-250 mmhg depending on size of person) or no blood flow restriction (placebo inflation) on right limb.

  * Protocol: 30 repetitions - 15 repetitions - 15 repetitions - 15 repetitions with each set separated by ~30-90 seconds.
  * Right and left legs will be alternating, but only one leg will have the occlusion cuff

Session 14 - Re-test

- Re-check 1RM, isometric quad strength, as well as muscle thickness of quadriceps with ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49

Exclusion Criteria:

* Pregnant
* Hypertensive
* Recent back or lower extremity injury
* History of blood clotting
* Varicose veins
* Adults lacking the capacity to consent for themselves

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Schoenecker, DPT, Principal Investigator — Fairview Health Services
Locations (1):
- Fairview Health Services, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Research coordinator/statistician will have access to blinded, individual data for the purpose of record keeping and analysis.

REFERENCES:
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Slysz J, Stultz J, Burr JF. The efficacy of blood flow restricted exercise: A systematic review & meta-analysis. J Sci Med Sport. 2016 Aug;19(8):669-75. doi: 10.1016/j.jsams.2015.09.005. Epub 2015 Sep 28. PMID 26463594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Flow Restriction Cuff | Blood Flow Restriction Cuff-Placebo
Started | 8 | 0
Completed | 7 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants completed the placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Flow Restriction Cuff | Blood Flow Restriction Cuff-Placebo | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.2) |  | 28.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8
One Repetition Maximum [Mean (Standard Deviation); unit: pounds] — Population: 8 participants were enrolled. 1 participants dropped-out prior to collection of this data measure.
  pounds
    number analyzed (Participants) | 7 | 0 | 7
    (all) | 267.1 (63.2) |  | 267.1 (63.2)
Quadriceps Muscle Thickness [Mean (Standard Deviation); unit: centimeters] — Population: 8 participants were enrolled. 1 participants dropped-out prior to collection of this data measure.
  centimeters
    number analyzed (Participants) | 7 | 0 | 7
    (all) | 42.4 (10.2) |  | 42.4 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: One Repetition Maximum
Description: One repetition maximum on the single leg press. Isometric quadriceps extension strength.
Time Frame: 6 weeks
Population: No participants completed the placebo arm.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Blood Flow Restriction Cuff | Blood Flow Restriction Cuff-Placebo
Number analyzed (Participants) | 7 | 0
pounds | 302.9 (67.1) |

2. Secondary Outcome: Quadriceps Muscle Thickness
Description: Difference between groups in the measurement of the muscle thickness of the quadriceps muscle via ultrasound.
Time Frame: 6 weeks
Population: No participants completed the placebo arm.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Blood Flow Restriction Cuff | Blood Flow Restriction Cuff-Placebo
Number analyzed (Participants) | 7 | 0
centimeters | 45 (13.4) |

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: No participants completed the placebo arm.
Arm/Group | Blood Flow Restriction Cuff | Blood Flow Restriction Cuff-Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03055260/Prot_SAP_000.pdf